CLINICAL TRIAL: NCT05457712
Title: Nutrition In Preoperative Pediatric Congenital Heart Disease: A Randomized Clinical Trial
Brief Title: Nutrition In Preoperative Pediatric Congenital Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Irmandade Santa Casa de Misericórdia de Porto Alegre (Other); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Fernanda Lucchese, PHD, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5516-18
Record Dates: First submitted 2022-03-18; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Congenital Heart Defects; Underweight
Keywords: Heart Defects, Congenital; Infant; Preoperative Care; Nutritional Support
MeSH Terms: conditions — Heart Defects, Congenital; Thinness | interventions — Clinical Protocols

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, pragmatic, with blind evaluation of outcomes.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, full blinding will not be possible. However, the statistical analysis team will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In the first evaluation and after the patient's consent, a standardized complementary questionnaire will be applied, with demographic and clinical information. The nutritionist will carry out the anthropometric assessment, questionnaires and application of the protocol for this group. The energy and protein value of the prescribed diet will be followed according to the original protocol considering plans A, B or C, via a hypercaloric formula with a caloric density of 1kcal/ ml for infants starting 60 days preoperatively. The return for nutritional monitoring will take place after evaluation: weekly, biweekly or monthly.
  Interventions: Dietary Supplement: protocol
- Control group (Other): In the first evaluation and after the patient's consent, a standardized complementary questionnaire will be applied, with demographic and clinical information. The nutritionist will carry out the anthropometric assessment and questionnaires. Afterwards, they will be evaluated through the standard nutritional protocol of the nutrition clinic of the Institute of Cardiology and Children's Hospital Santo Antonio of Porto Alegre, whose standard nutritional prescription is a polymeric formula with a caloric density of 0.67 kcal/ml. Nutritional monitoring will take place through telephone contact for information on the baby's clinical data and in person before the surgery is performed.
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: protocol — The energy and protein value of the prescribed diet will be followed according to the original protocol considering plans A, B or C, via a hypercaloric formula with a caloric density of 1kcal/ml for infants starting 60 days preoperatively. The return for nutritional monitoring will take place after evaluation: weekly, biweekly or monthly.
  Arms: Intervention group
Other: Control — Afterwards, they will be evaluated through the standard nutritional protocol of the nutrition clinic of the Instituto de Cardiologia de and Hospital Santo Antonio de Porto Alegre, whose standard nutritional prescription is a polymeric formula with a caloric density of 0.67 kcal/ml. Nutritional monitoring will take place through telephone contact for information on the baby's clinical data and in person before the surgery is performed.
  Arms: Control group

SUMMARY:
Introduction: The use of a nutritional protocols provides the standardization of assessment procedures and the optimization of nutritional status recovery of pre-surgical infants with Congenital Heart Disease (CHD). However, to our knowledge there are no validated instrument for presurgical nutritional support for infants with congenital heart disease (CHD) in Brazil.

Objective: Assess the clinical effectiveness of the translated and cross-culturally adapted protocol, Nutritional Pathway for Infants with Congenital Heart Disease before Surgery (Marino et al., 2018), on the weight change of infants with congenital heart disease in two specialized cardiology hospitals in Southern Brazil in partnership with the UK research group that authored the original of protocol.

Methods: A randomized, pragmatic clinical trial will be carried out. The sample will consist of children with CHD, between 0-12 months of age, awaiting cardiovascular corrective surgery from the Pediatric Outpatient Clinic in the Institute of Cardiology (IC) and Children's Hospital Santo Antonio of Santa Casa de Misericordia. The previously translated pre-surgical nutritional intervention protocol for infants with congenital heart disease will be compared with current routine nutritional guidelines used in the follow-up services of children with congenital heart disease in these institutions within the national public healthcare, SUS.

Intended results: It is expected that the culturally-adapted pre-surgical nutritional support protocol for children with congenital heart disease will be effective in pre-surgical infant weight gain, which will likely improve surgical prognosis and clinical outcomes. And we hope that this protocol will promote the standardization of care, and will provide an empirically-based nutritional intervention that may improve the effectiveness of nutritional recovery in the CHD infants. Furthermore, the results may be used in the formulation of Brazilian guidelines for comprehensive care of children with congenital heart disease.

DETAILED DESCRIPTION:
OBJECTIVES

* Test the clinical effectiveness of the translation and adaptation of a pre-surgical nutritional intervention protocol for children with CHD on pre-surgical weight gain, as well as, compare it with the current clinical practice in Brazil.
* Assess the nutritional status of the participants;

A NUTRITIONAL PROTOCOL IN PRE-SURGICAL PEDIATRIC CONGENITAL HEART DISEASE IN BRAZIL: A RANDOMIZED PRAGMATIC CLINICAL TRIAL

DESIGN Randomized clinical trial, pragmatic, blinded for outcomes evaluation. Following the Consolidated Standards of Reporting Trials (CONSORT) guidelines for the writing of randomized clinical trials.

POPULATION The population from which the sample will be randomized will consist of children with congenital heart disease, aged from 0-12 months, in the pre-operative phase and from the Pediatrics Clinic of the Institute of Cardiology (IC), and Children's Hospital Santo Antonio, located in the city of Porto Alegre, RS, Brazil.

STUDY LOGISTICS Patients will be referred to the pediatric outpatient clinic of the Institute of Cardiology (IC) of Porto Alegre and/or the pediatric outpatient clinic of the Children's Hospital Santo Antonio by the accompanying physician according to pre-established eligibility criteria. The caregivers will be invited to participate in the study. The electronic Consent Form link will be sent to the person responsible, which he/she should read, resolve doubts with the team, and only then digitally sign accepting to participate in the study. After signing the consent form, an appointment will be scheduled to be held at the institution' pediatric outpatient clinics, where the methodology, study objectives and randomization to the control or intervention group will be explained.

STUDY VARIABLES: DEMOGRAPHIC AND CLINICAL To obtain the baseline data, a structured questionnaire developed for this research will be used, which will include social, biological and demographic data. Among the clinical data, information regarding the diagnosis of CHD, food intake and feeding routine, swallowing difficulties, previous hospitalizations, comorbidities, medications in use, and anthropometric data will be collected.

Hypothesis:

Using a specific nutritional protocol for infants with pre-surgical congenital heart disease can minimize growth/weight deficits and improve post-surgical prognosis.

STUDY INTERVENTION

Intervention group In the first evaluation and after the patient's consent, a standardized complementary questionnaire will be applied, with demographic and clinical information. The nutritionist will carry out the anthropometric assessment, questionnaires and application of the protocol for this group. The measurements will be determined with the aid of a digital Filizola® pediatric scale, duly calibrated, with a maximum value of 15kg and 5g division. To measure the head circumference, a measuring tape graduated in non-elastic millimeters will be used, and a child anthropometer will be used to measure height. The steps of the protocol to be translated using the criteria will be used: assess the nutritional risk according to the type of cardiac injury (with higher risk those children who present more than one type of congenital injury or more severe); monitor growth through weight, length and head circumference; assess feeding skills as well as lack of progress or regression from previous skills; assess food intake, whether adequate or not for weight gain; determine which nutritional care plan is appropriate based on any prior assessment. The energy and protein value of the prescribed diet will be followed according to the original protocol considering plans A, B or C, via a hypercaloric formula with a caloric density of 1kcal/ml for infants starting 60 days preoperatively. The return for nutritional monitoring will take place after evaluation: weekly, biweekly or monthly.

Control group In the first evaluation and after the patient's consent, a standardized complementary questionnaire will be applied, with demographic and clinical information. The nutritionist will carry out the anthropometric assessment and questionnaires. Afterwards, they will be evaluated through the standard nutritional protocol of the nutrition clinic of the IC and SACH whose standard nutritional prescription is a polymeric formula with a caloric density of 0.67 kcal/ml.

Nutritional monitoring will take place through telephone contact for information on the baby's clinical data and in person before the surgery is performed.

ETHICAL CONSIDERATIONS The Project is already approved by the Research Ethics Committee of the Institute of Cardiology - University Foundation of Cardiology, Porto Alegre - RS, under number 5516/18. It was presented and approved by the cardiology team of the Hospital Sao Francisco and approved by the CEP of the Children's Hospital Santo Antonio da Santa Casa de Misericordia in Porto Alegre.

Those responsible for the children who will participate in the research must sign a TCLE, as well as the members of the expert committee of which they will retain a copy, being guaranteed by the study team that the ethical principles of the research in human beings provided for in Resolution 466/2012 of 12/12/2012 of the National Health Council will be respected.

ELIGIBILITY:
Inclusion Criteria:

* Children with a diagnosis of congenital heart disease aged between zero and twelve months, awaiting surgery for cardiac correction, classified in risk category 1 of the RACHS-1 score;
* Term birth;

Exclusion Criteria:

* Patients with:

  * Neurological impairment;
  * Craniofacial malformation;
  * Structural alterations of the upper airways;
  * Respiratory impairment;
  * Suspicion or diagnosis of genetic syndrome;
  * Any type of food allergy.

Ages: 30 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Estimated)
Dates: Start 2023-01-09 (Estimated); Primary Completion 2024-04-02 (Estimated); Study Completion 2024-05-02 (Estimated)

PRIMARY OUTCOMES:
changing the nutritional status | change in nutritional status after 60 days of preoperative intervention
  Effectiveness of the cross-culturally adapted protocol on changing the nutritional status of babies with congenital heart disease

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Lucchese, PhD, Principal Investigator — Instituto de Cardiologia do Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marino LV, Johnson MJ, Hall NJ, Davies NJ, Kidd CS, Daniels ML, Robinson JE, Richens T, Bharucha T, Darlington AE; British Dietetic Association Paediatric Cardiology Interest Group. The development of a consensus-based nutritional pathway for infants with CHD before surgery using a modified Delphi process. Cardiol Young. 2018 Jul;28(7):938-948. doi: 10.1017/S1047951118000549. Epub 2018 Apr 29. PMID 29704905
- See also: The development of a consensus-based nutritional pathway for infants with CHD before surgery using a modified Delphi process — https://pubmed.ncbi.nlm.nih.gov/29704905/